CLINICAL TRIAL: NCT07269743
Title: To OBSERVE PRACTISE OF AEROSOL THERAPY IN ARDS PATIENTS (AERO-IN-ARDS)
Brief Title: AEROSOL THERAPY IN ARDS PATIENTS (AERO-IN-ARDS)
Acronym: AERO-IN-ARDS
Status: Recruiting | Type: Observational
Sponsor: TS Misra Medical College (Other)
Collaborators: All India Institute of Medical Sciences (Other); All India Institute of Medical Sciences, Raipur (Other Government); Ram Manohar Lohia Institute of Medical Sciences, Lucknow (Unknown); Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government); Hospital General Universitario Morales Meseguer (Other); Istanbul Medipol University Hospital (Other); Casa di Cura del Policlinico di Milano (Unknown); HOSPITAL BRITANICO DE BUENOS AIRES (Other)
Responsible Party: Principal Investigator, PIYUSH SRIVASTAVA, DR PIYUSH SRIVASTAVA, TS Misra Medical College
Other Study IDs: TSMMC-2025-237(6)
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome) Receiving IMV
Keywords: ARDS; AEROSOL THERAPY; INVASIVE MECHANICAL VENTILATION
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ARDS PATIENTS: REQUIREING INVASIVE MECHANICAL VENTILATION
  Interventions: Drug: Types of drugs being delivered as aerosol therapy

INTERVENTIONS:
Drug: Types of drugs being delivered as aerosol therapy — Every time the patient receives inhaled medication, except for the instillation of 0.9% normal saline in the artificial airway for suctioning, will be counted in aerosol therapy.

SUMMARY:
Aerosol therapy delivers medicines as a fine mist directly into the lungs. This allows faster action and fewer whole-body side effects. It is a key treatment for diseases such as asthma and COPD. In acute respiratory distress syndrome (ARDS), early laboratory and small clinical studies suggested that inhaled beta-2 agonists and corticosteroids might help the lungs heal by improving mucus clearance, reducing inflammation, and helping remove excess fluid. However, larger randomized trials have not shown clear clinical benefits. Therefore, major guidelines do not provide specific recommendations for aerosol use in ARDS. There are also safety concerns, including risks of low potassium levels, abnormal heart rhythms, worsening lung function, and increased healthcare costs. Despite these uncertainties, our previous study showed that aerosol therapy continues to be used widely in ARDS patients. However, that study was small and limited to one country, so the findings may not apply to other regions.

To address this gap, we have designed Aero-in-ARDS, a large, multi-national, prospective observational study. This study will investigate how often aerosol therapy is used in ARDS, what types of aerosol drugs are given, and how practices differ across countries. By identifying current patterns and comparing them with existing evidence, the study aims to highlight gaps in knowledge and guide future research.

DETAILED DESCRIPTION:
This prospective, multi-center, international cohort observational study will be conducted upon approval from the Institutional Ethics Committee (IEC). Centers' recruitment from various parts of the Globe will be done on an invitation basis. Participation in centers will be purely voluntary. As per their local policy, the participating center will take additional IEC approval or waiver at their center to initiate enrollment. Requests for patients' or legal representatives' informed consent will be made in accordance with national law.

The study protocol is designed and will be reported in accordance with the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement. All consecutive eligible patients with ARDS admitted to participating ICUs will be enrolled. The study aims to include all consecutive eligible patients to ensure accurate and representative data collection. Each Participating center will screen all consecutive ARDS patients requiring invasive mechanical ventilation during the study's six-month inclusion period, or a maximum of 25 patients per center. Patients who met the inclusion/exclusion criteria will be followed for the next 14 days or till ICU discharge/death or weaning from IMV, whichever comes first.

ELIGIBILITY:
Inclusion Criteria: all newly admitted adult patients with a diagnosis of ARDS in the participating ICU

1. The patient requires mechanical ventilation.
2. Age ≥ 18 years
3. Informed consent (if required)

Exclusion Criteria:

1. Age <18 years
2. Patients managed with NIV, and HFNO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each Participating center will screen all consecutive ARDS patients requiring invasive mechanical ventilation during the study's six-month inclusion period, or a maximum of 25 patients per center. Patients who met the inclusion/exclusion criteria will be followed for the next 14 days or till ICU discharge/death or weaning from IMV, whichever comes first.
Sampling Method: Non-Probability Sample
Enrollment: 423 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
FREQUENCY OF AEROSOL THERAPY | 6 MONTHS
  HOW MANY ARDS PATIENTS WERE RECEIVING AEROSOL THERAPY
TYPES OF drug USED as aerosol therapy | 6 MONTHS
  HOW MANY TYPES OF DRUGS WERE USED AS AEROSOL THERAPY IN ARDS PATIENTS
frequency of aerosol therapy | 6 MONTHS
  FREQUENCY OF AEROSOL THERAPY IN ARDS PATIENTS ON IMV
types of drugs use as aerosol therapy | 6 months
  types of drugs use as aerosol therapy in ARDS patients while receiving Invasive Mechanical Ventilation

SECONDARY OUTCOMES:
Modality used for aerosol drug delivery | 6 MONTHS
  TYPES OF AEROSOL GENERATORS USED TO DELIVER AEROSOL THERAPY IN ARDS PATIENTS
Types of aerosol generators used for aerosol drug delivery | 6 months
  Types of aerosol generators used for aerosol drug delivery in ARDS patients while receiving IMV

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Gurjjar, MD, Study Chair — SGPGIMS; Berkan Basancelebi, RT, PT, MSc, FNIV, Study Chair — Medipol University; Gustavo Plotnikow, BPT, BCs, PhD(c), Study Chair — Servicio de Rehabilitación, área de Kinesiología UCI, Hospital Británico de Buenos Aires, Buenos Aires, Argentina Facultad de Medicina Y Ciencias de la Salud, Universidad Abierta lnteramericana, Buenos Aires, Argentina; Giuseppe Francesco Sferrazza Papa, MD PhD, Study Chair — Casa di cura policlinico, department of rehabilitation sciences, Milan, (Italy); Salvatore Notaro, MD, Study Chair — AORN colli Hospitals; Antonio M Esquinas, MD, PhD, FCCP, FNIV, FBCV, Study Chair — Instituto Murciano de Investigacion Biosanitaria, Murcia, Spain
Locations (1):
- Ts Misra Medical College, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
Access to STUDY IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after publication of manuscript and the data will be made accessible for up to 24 months
Access Criteria: qualified researchers engaging in independent scientific research

REFERENCES:
- [Background] Singhal S, Saran S, Joshi K, Gurjar M, Rao PB, Sahoo JN, Dua R, Sahoo AK, Sharma A, Agarwal S, Sharma A, Ghosh PS, Kothari N, Deokar K, Mukherjee S, Sharma P, Sreedevi B, Sivaramakrishnan P, Singh U, Sundaram D, Agrawal A. Practice pattern of aerosol drug therapy in ARDS patients: A secondary analysis of the Aero-in-ICU study. J Intensive Med. 2025 Jul 5;5(4):385-391. doi: 10.1016/j.jointm.2025.05.003. eCollection 2025 Oct. PMID 41180103
- [Background] Singhal S, Gurjar M, Sahoo JN, Saran S, Dua R, Sahoo AK, Sharma A, Agarwal S, Sharma A, Ghosh PS, Rao PB, Kothari N, Joshi K, Deokar K, Mukherjee S, Sharma P, Sreedevi BP, Sivaramakrishnan P, Singh U, Sundaram D, Agrawal A, Katoch CDS. Aerosol drug therapy in critically ill patients (Aero-in-ICU study): A multicentre prospective observational cohort study. Lung India. 2024 May 1;41(3):200-208. doi: 10.4103/lungindia.lungindia_580_23. Epub 2024 Apr 30. PMID 38687231